CLINICAL TRIAL: NCT05504148
Title: Protection of Cardiovascular Function With Crocin in BrEast Cancer Patients Undergoing Radiotherapy and Chemotherapy
Acronym: ProtECtion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6010121027
Record Dates: First submitted 2022-08-04; First posted 2022-08-17 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Cancer therapy-related cardiac dysfunction; Crocin; Echocardiography; Speckle tracking technology
MeSH Terms: conditions — Breast Neoplasms | interventions — crocin

STUDY DESIGN:
Intervention Model Description: Inclusion criteria:
  1. Age 25-80 years old, female;
  2. Patients diagnosed with breast cancer by histopathology;
  3. Patients who plan to receive adjuvant radiotherapy/chemotherapy or combined adjuvant trastuzumab or pertuzumab targeted therapy;
  4. Patients who completed at least 6 cycles of treatment after enrollment;
  Exclusion criteria:
  1. pregnant or breastfeeding women;
  2. Patients with poor echocardiographic image quality;
  3. Persistent atrial fibrillation and severe arrhythmia affect the collection and analysis of ultrasound data;
  4. Patients who are participating in other clinical studies.
  Eligible patients were randomly divided into 1:1 group and divided into crocin group and placebo control group. Both groups of subjects received crocin or placebo on the basis of standard anti-tumor treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crocin group (Experimental): The chemotherapy/radiotherapy protocols are made by oncologists adopted for patients depending on specific conditions , take saffron total glucosides tablets(provided by Reyoung Pharmaceutical Co., Ltd.) for 8 days during each chemotherapy (started on the 1st day before chemotherapy), 4 tablets/time, 3 times a day.
  Interventions: Drug: crocin
- placebo group (Placebo Comparator): Undergoing chemotherapy/radiotherapy protocols as planned, take placebo piece during(the same appearance of crocin tablets, production unit:Reyoung Pharmaceutical Co., Ltd.) for 8 days during each chemotherapy (started on the 1st day before chemotherapy), 4 tablets/time, 3 times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: crocin — Take saffron total glucosides tablets for 8 days during each chemotherapy (started on the 1st day before radiotherapy/chemotherapy), 4 tablets/time, 3 times a day.
  Arms: Crocin group
Drug: Placebo — Take placebo piece during for 8 days during each chemotherapy (started on the 1st day before radiotherapy/chemotherapy), 4 tablets/time, 3 times a day
  Arms: placebo group

SUMMARY:
The potential cardiovascular toxicity of tumor treatment and its resulting cardiovascular events have gradually become an important health risk for tumor survivors. Prevention and early identification of cardiovascular toxicity has now become one of the bottlenecks in improving the prognosis of cancer patients. Compared to conventional echocardiographic indicators, new ultrasound technology based on speckle tracking imaging (STI) has shown superiority in the diagnosis, risk stratification and prognosis evaluation of cardiovascular diseases. Crocin, one of the main active components of saffron, has been found protective effect on cardiovascular toxicity in basic studies. This is a randomized, double-blind, placebo-controlled, single-center clinical study to observe the effect of crocin on cardiovascular function caused by breast cancer treatment.

One hundred and twenty breast cancer patients planning to undergo radiotherapy or chemotherapy will be included and randomly divided into a crocin group and a placebo group to observe the effect of total saffron tablets on cardiovascular function in patients with early breast cancer radiotherapy and chemotherapy. Participants will take crocin or placebo (4 tablets/time, 3 times a day) during each cycle of chemotherapy for 8 days, started on the 1st day before radiotherapy/chemotherapy. Follow-up was performed every 3 months after enrollment, and the follow-up period was 6 months.

Primary study endpoints include the differences between groups in the difference in LVEF and GLS measured by echocardiography at the end of the experiment compared to baseline. Secondary study endpoint include the differences in the incidence rates of serum troponin exceeding the upper limit of normal value and NT-proBNP higher than the normal age reference value, the frequency and duration of chest tightness, chest pain and palpitation, the degree of arrhythmia and ST-T changes displayed by dynamic electrocardiogram, the other echocardiographic parameters (the E/e', global circumferential strain, global radial strain, 3D-GAS, LV torsion, LV rotation/derotation velocity, SDI, RVFWS, and indexes of left ventricular diastolic function and right ventricular function) at the end of the experiment compared to baseline between the two groups.

ELIGIBILITY:
Inclusion criteria:

1. Age 25-80 years old, female;
2. Patients diagnosed with breast cancer by histopathology;
3. Patients who plan to receive adjuvant radiotherapy/chemotherapy or combined adjuvant trastuzumab or pertuzumab targeted therapy;
4. Patients who completed at least 6 cycles of treatment after enrollment;

Exclusion criteria:

1. pregnant or breastfeeding women;
2. Patients with poor echocardiographic image quality;
3. Persistent atrial fibrillation and severe arrhythmia affect the collection and analysis of ultrasound data;
4. Patients who are participating in other clinical studies.

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-09-25 (Estimated)

PRIMARY OUTCOMES:
The change of LVEF measured by echocardiography | At the end of 6-month follow-up compared to the baseline
  The differences between the two groups in the difference of LVEF measured by Echocardiography at the end of the experiment compared to that at the baseline.
The change of GLS measured by echocardiography | At the end of 6-month follow-up compared to the baseline
  The differences between the two groups in the difference of GLS measured by Echocardiography at the end of the experiment compared to that at the baseline.

SECONDARY OUTCOMES:
The incidences of the increase of serum troponin and/or NT-proBNP | During 6 months of following up
  Differences in the incidence rates of serum troponin exceeding the upper limit of normal value and NT-proBNP higher than the normal age reference value between the two groups during follow-up.
The incidences of chest tightness, chest pain and palpitation | During 6 months of following up
  The differences in the incidence of chest tightness, chest pain and palpitation between the two groups
The incidences of arrhythmia and ST-T changes | During 6 months of following up
  Differences between the two groups in the incidences of arrhythmia and ST-T changes displayed by dynamic electrocardiogram.
The differences of global circumferential strain, global radial strain, global area strain measured by echocardiography. | At the end of 6-month follow-up compared to the baseline
  Differences between groups in the difference in global circumferential strain, global radial strain, global area strain measured by echocardiography at the end of the experiment compared to baseline.
The indexes of E, e', a', tricuspid regurgitation velocity measured by echocardiography. | At the end of 6-month follow-up compared to the baseline
  Differences between groups in the difference in the indexes of left ventricular diastolic function measured by echocardiography at the end of the experiment compared to baseline.
The indexe of E/e'measured by echocardiography. | At the end of 6-month follow-up compared to the baseline
  Differences between groups in the difference in the indexes of left ventricular diastolic function measured by echocardiography at the end of the experiment compared to baseline.
The indexe of left atrial volume index (LAVI)measured by echocardiography. | At the end of 6-month follow-up compared to the baseline
  Differences between groups in the difference in the indexes of left ventricular diastolic function measured by echocardiography at the end of the experiment compared to baseline.
The indexe of TAPSE measured by echocardiography. | At the end of 6-month follow-up compared to the baseline
  Differences between groups in the difference in the right ventricular function monitoring indicators measured by echocardiography at the end of the experiment compared to baseline.
The indexe of RV fractional area change (FAC) measured by echocardiography. | At the end of 6-month follow-up compared to the baseline
  Differences between groups in the difference in the right ventricular function monitoring indicators measured by echocardiography at the end of the experiment compared to baseline.
The indexe of right ventricular free wall global longitudinal strain (RVGLS) measured by echocardiography. | At the end of 6-month follow-up compared to the baseline
  Differences between groups in the difference in the right ventricular function monitoring indicators measured by echocardiography at the end of the experiment compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Zhang, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the study protocol,statistical Analysis Plan (SAP)and Informed Consent Form (ICF)of this research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The sharing time period is 6 months to 1 year after the data is released.
Access Criteria: Share IPD under the conditions of protecting the privacy of patients and ensuring the safety of all diseases.
  It is necessary to contact the researcher and open the sharing authority after the researcher's consent.

REFERENCES:
- [Background] Zamorano JL, Lancellotti P, Rodriguez Munoz D, Aboyans V, Asteggiano R, Galderisi M, Habib G, Lenihan DJ, Lip GYH, Lyon AR, Lopez Fernandez T, Mohty D, Piepoli MF, Tamargo J, Torbicki A, Suter TM; ESC Scientific Document Group. 2016 ESC Position Paper on cancer treatments and cardiovascular toxicity developed under the auspices of the ESC Committee for Practice Guidelines: The Task Force for cancer treatments and cardiovascular toxicity of the European Society of Cardiology (ESC). Eur Heart J. 2016 Sep 21;37(36):2768-2801. doi: 10.1093/eurheartj/ehw211. Epub 2016 Aug 26. No abstract available. PMID 27567406
- [Background] Tarantini L, Gulizia MM, Di Lenarda A, Maurea N, Giuseppe Abrignani M, Bisceglia I, Bovelli D, De Gennaro L, Del Sindaco D, Macera F, Parrini I, Radini D, Russo G, Beatrice Scardovi A, Inno A. ANMCO/AIOM/AICO Consensus Document on clinical and management pathways of cardio-oncology: executive summary. Eur Heart J Suppl. 2017 May;19(Suppl D):D370-D379. doi: 10.1093/eurheartj/sux019. Epub 2017 May 2. PMID 28751851
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Arai M, Tomaru K, Takizawa T, Sekiguchi K, Yokoyama T, Suzuki T, Nagai R. Sarcoplasmic reticulum genes are selectively down-regulated in cardiomyopathy produced by doxorubicin in rabbits. J Mol Cell Cardiol. 1998 Feb;30(2):243-54. doi: 10.1006/jmcc.1997.0588. PMID 9515001
- [Background] Papadopoulou LC, Theophilidis G, Thomopoulos GN, Tsiftsoglou AS. Structural and functional impairment of mitochondria in adriamycin-induced cardiomyopathy in mice: suppression of cytochrome c oxidase II gene expression. Biochem Pharmacol. 1999 Mar 1;57(5):481-9. doi: 10.1016/s0006-2952(98)00305-0. PMID 9952311
- [Background] Chen XL, Lei YH, Liu CF, Yang QF, Zuo PY, Liu CY, Chen CZ, Liu YW. Angiogenesis inhibitor bevacizumab increases the risk of ischemic heart disease associated with chemotherapy: a meta-analysis. PLoS One. 2013 Jun 20;8(6):e66721. doi: 10.1371/journal.pone.0066721. Print 2013. PMID 23818962
- [Background] Schutz FAB, Je Y, Azzi GR, Nguyen PL, Choueiri TK. Bevacizumab increases the risk of arterial ischemia: a large study in cancer patients with a focus on different subgroup outcomes. Ann Oncol. 2011 Jun;22(6):1404-1412. doi: 10.1093/annonc/mdq587. Epub 2010 Nov 29. PMID 21115602
- [Background] Ranpura V, Hapani S, Chuang J, Wu S. Risk of cardiac ischemia and arterial thromboembolic events with the angiogenesis inhibitor bevacizumab in cancer patients: a meta-analysis of randomized controlled trials. Acta Oncol. 2010 Apr;49(3):287-97. doi: 10.3109/02841860903524396. PMID 20156114
- [Background] Suter TM, Ewer MS. Cancer drugs and the heart: importance and management. Eur Heart J. 2013 Apr;34(15):1102-11. doi: 10.1093/eurheartj/ehs181. Epub 2012 Jul 12. PMID 22789916
- [Background] Carver JR, Shapiro CL, Ng A, Jacobs L, Schwartz C, Virgo KS, Hagerty KL, Somerfield MR, Vaughn DJ; ASCO Cancer Survivorship Expert Panel. American Society of Clinical Oncology clinical evidence review on the ongoing care of adult cancer survivors: cardiac and pulmonary late effects. J Clin Oncol. 2007 Sep 1;25(25):3991-4008. doi: 10.1200/JCO.2007.10.9777. Epub 2007 Jun 18. PMID 17577017
- [Background] Malanca M, Cimadevilla C, Brochet E, Iung B, Vahanian A, Messika-Zeitoun D. Radiotherapy-induced mitral stenosis: a three-dimensional perspective. J Am Soc Echocardiogr. 2010 Jan;23(1):108.e1-2. doi: 10.1016/j.echo.2009.08.006. Epub 2009 Sep 18. PMID 19766451
- [Background] Darby SC, Cutter DJ, Boerma M, Constine LS, Fajardo LF, Kodama K, Mabuchi K, Marks LB, Mettler FA, Pierce LJ, Trott KR, Yeh ET, Shore RE. Radiation-related heart disease: current knowledge and future prospects. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):656-65. doi: 10.1016/j.ijrobp.2009.09.064. PMID 20159360
- [Background] Plana JC, Galderisi M, Barac A, Ewer MS, Ky B, Scherrer-Crosbie M, Ganame J, Sebag IA, Agler DA, Badano LP, Banchs J, Cardinale D, Carver J, Cerqueira M, DeCara JM, Edvardsen T, Flamm SD, Force T, Griffin BP, Jerusalem G, Liu JE, Magalhaes A, Marwick T, Sanchez LY, Sicari R, Villarraga HR, Lancellotti P. Expert consensus for multimodality imaging evaluation of adult patients during and after cancer therapy: a report from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2014 Oct;15(10):1063-93. doi: 10.1093/ehjci/jeu192. No abstract available. PMID 25239940
- [Background] Amundsen BH, Helle-Valle T, Edvardsen T, Torp H, Crosby J, Lyseggen E, Stoylen A, Ihlen H, Lima JA, Smiseth OA, Slordahl SA. Noninvasive myocardial strain measurement by speckle tracking echocardiography: validation against sonomicrometry and tagged magnetic resonance imaging. J Am Coll Cardiol. 2006 Feb 21;47(4):789-93. doi: 10.1016/j.jacc.2005.10.040. Epub 2006 Jan 26. PMID 16487846
- [Background] Huang SJ, Orde S. From speckle tracking echocardiography to torsion: research tool today, clinical practice tomorrow. Curr Opin Crit Care. 2013 Jun;19(3):250-7. doi: 10.1097/MCC.0b013e32836092b7. PMID 23519081
- [Background] Razmaraii N, Babaei H, Mohajjel Nayebi A, Assadnassab G, Ashrafi Helan J, Azarmi Y. Crocin treatment prevents doxorubicin-induced cardiotoxicity in rats. Life Sci. 2016 Jul 15;157:145-151. doi: 10.1016/j.lfs.2016.06.012. Epub 2016 Jun 11. PMID 27297631
- [Background] Razavi BM, Hosseinzadeh H, Movassaghi AR, Imenshahidi M, Abnous K. Protective effect of crocin on diazinon induced cardiotoxicity in rats in subchronic exposure. Chem Biol Interact. 2013 May 25;203(3):547-55. doi: 10.1016/j.cbi.2013.03.010. Epub 2013 Mar 21. PMID 23523949

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT05504148/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT05504148/ICF_001.pdf